CLINICAL TRIAL: NCT03452735
Title: Fertility Study of Women With Chronic Inflammatory Rheumatism
Acronym: FERTIRHUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0446; 2017-A03539-44 (Other: ID-RCB)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Arthritis, Psoriatic; Arthritis, Rheumatoid; Ankylosing Spondylitis; Chronic Juvenile Arthritis
Keywords: Chronic inflammatory rheumatism; Fertility; Procreation
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients diagnosed before age 40: Patient between 18 and 50 years-old with Rheumatoid arthritis, Psoriatic arthritis, Ankylosing spondylitis, Chronic juvenile arthritis, Chronic Inflammatory Rheumatism who will answer to a questionnaire about fertility
  Interventions: Other: Questionnaire about fertility
- Control Group: Patient between the ages of 18 and 50 years, not diagnosed with Chronic inflammatory rheumatism, having consulted in Rheumatology for a mechanical pathology, presenting no chronic pathology, having no chemo or radiotherapy or immunosuppressive therapy, or pelvic surgery before age 40 years who will answer to a questionnaire about fertility
  Interventions: Other: Questionnaire about fertility

INTERVENTIONS:
Other: Questionnaire about fertility — Sending a questionnaire about fertility that will have to be returned to us in order to be included in the study. The questionnaires, anonymous, will be numbered according to their order of return.

SUMMARY:
Etiopathogenesis of Chronic inflammatory rheumatisms (CIR) includes genetic, autoimmune and environmental factors. Their impact on the quality of life is important, leading to a sometimes severe disability. Thus they are likely to affect female fertility through several mechanisms, including autoimmune since the association between immunity and fertility has already been demonstrated in other autoimmune diseases.

This study wants to evaluate and compare the birth rate between CIR and control group.

DETAILED DESCRIPTION:
Data collection will be carried out using a questionnaire submitted to women in charge of the rheumatology department of the University Hospital of Toulouse and having agreed to participate:

* women with Rheumatoid arthritis, Psoriatic arthritis, Ankylosing spondylitis or Chronic juvenile arthritis for the chronic inflammatory rheumatism group
* women with a mechanical rheumatic pathology for the control group

The primary endpoint was birth rate after spontaneous or induced pregnancy in patients who attempted to procreate, in the CIR group and in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Rheumatoid arthritis, Psoriatic arthritis, Ankylosing spondylitis, Chronic juvenile arthritis, Chronic Inflammatory Rheumatism
* Patient diagnosed before the age of 40
* Patient having given her no opposition to her participation in research
* For the control group: patient not suffering from chronic inflammatory rheumatism, having consulted in Rheumatology for a mechanical pathology

Exclusion Criteria:

* Patient> 40 years old at the time of diagnosis
* Patient with insufficient medical data (treatments)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — study on woman fertility
Study Population: * Case group: patient with Rheumatoid arthritis, Psoriatic arthritis, Ankylosing spondylitis, Chronic juvenile arthritis
  * Control Group: patient not suffering from RIC, having consulted in rheumatology for a mechanical pathology (eg osteoarthritis, mechanical low back pain ...)
Sampling Method: Non-Probability Sample
Enrollment: 2900 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Birth rate after spontaneous or induced pregnancy | One day
  Birth rate after spontaneous or induced pregnancy in women who have tried to procreate in the chronic inflammatory rheumatism group and in the control group.

SECONDARY OUTCOMES:
Rates of ectopic pregnancy, early or late spontaneous miscarriage | one day
  Rates of ectopic pregnancy, early or late spontaneous miscarriage, early or late pregnancy, children born dead, preterm birth in the CIR group and in the control group
Design time | One day
  Design time in the CIR group and in the control group
Birth rate according to the treatments used | One day
  Birth rate in the CIR group according to the treatments used
Birth rate according to the activity of the disease | One day
  Birth rate in the CIR group according to the activity of the disease
Rates of desire for pregnancy | One day
  Rates of desire for pregnancy and study of the reasons for this lack of desire for pregnancy in the CIR group and in the control group
Rates of sexual dysfunction | One day
  Rates of sexual dysfunction in the CIR group and in the control group

CONTACTS AND LOCATIONS:
Overall Officials: Jean Parinaud, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No